CLINICAL TRIAL: NCT06498973
Title: CD123 Antibody Toxin Congregate (CD123 ATC; Tagraxofusp) Combined With Azacitidine for Maintenance Therapy Post Allogeneic Hematopoietic Cell Transplantation for Patients With CD123-Positive Malignant
Brief Title: Tagraxofusp and Azacitidine for Maintenance Treatment in Patients With CD123 Positive AML and MDS Following Donor Hematopoietic Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23400; NCI-2024-05359 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23400 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Specimen Handling; Biopsy; tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tagraxofusp, azacitidine) (Experimental): Patients receive tagraxofusp IV over 15 minutes QD on days 1-3 and azacitidine IV over 10-40 minutes QD on days 1-5 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and bone marrow aspiration and biopsy on study.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Other: Questionnaire Administration; Biological: Tagraxofusp-erzs

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Other: Questionnaire Administration — Ancillary studies
Biological: Tagraxofusp-erzs — Given IV
  Other Names: Diphtheria Toxin(388)-Interleukin-3 Fusion Protein; DT(388)-IL3 Fusion Protein; DT388IL3 fusion protein; Elzonris; IL3R-targeting Fusion Protein SL-401; SL 401; SL-401; SL401; Tagraxofusp; Tagraxofusp ERZS

SUMMARY:
This phase Ib trial tests the safety, side effects, best dose and effectiveness of tagraxofusp in combination with azacitidine as maintenance therapy in treating patients with CD123 positive acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) after a donor (allogeneic) hematopoietic cell transplant. An allogeneic hematopoietic cell transplant (HCT) is a type of transplant where the cancer patient receives cells from another person. Maintenance therapy is given after the transplant to prevent the cancer from coming back. Tagraxofusp is a drug that targets cells that have CD123 on their surface in order to kill the cancer cells to help prevent the cancer from coming back. Azacitidine is in a class of medications called demethylation agents. It works by helping the bone marrow to produce normal blood cells and by killing abnormal cells. Giving tagraxofusp in combination with azacitidine may be safe, tolerable and/or effective maintenance therapy in patients with CD123 positive AML and MDS after an allogeneic HCT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety and feasibility of tagraxofusp-erzs (tagraxofusp) with a fixed dose of azacitidine and determine the recommended phase 2 dose (RP2D) for tagraxofusp in patients with CD123-positive hematological malignancy when given as maintenance therapy following allogeneic transplant (HCT).

SECONDARY OBJECTIVES:

I. Estimate overall survival (OS), progression-free survival (PFS) and the cumulative incidence of relapse and non-relapse mortality (NRM) at 100 days and 1 year after starting maintenance therapy.

II. Evaluate the cumulative incidence of grade 2-4 and 3-4 acute graft-versus-host disease (GVHD) at 100 days post-HCT, secondary graft failure, and chronic GVHD at 1-year after HCT.

III. Estimate the cumulative incidence of infections in the first 100 days from the start of maintenance therapy.

EXPLORATORY OBJECTIVES:

I. Describe kinetics of immune cell recovery during 1st year post-HCT and during maintenance therapy with tagraxofusp-azacitidine (TAG-AZA).

II. Assess the possible correlation between chimerism kinetics (per next generation sequencing [NGS]/ quantitative polymerase chain reaction [qPCR] assay) and post-HCT relapse during maintenance therapy with TAG-AZA.

III. Characterize the presence and level of GVHD biomarkers and inflammatory cytokines in the first 100 days from the start of maintenance therapy.

IV. Assess patients' quality of life (QOL) at baseline (before initiation of the first cycle) then at the end of cycles 3 and 6 (± 2 weeks); optional questionnaire.

V. Longitudinally assess CD123 expression on hematopoietic cells. VI. Assess changes in symptoms of chronic GVHD using Lee Symptom Scale; patient self-report.

VII. Describe transplant outcomes defined in the secondary objectives among all consented patients regardless of receiving the study therapy.

OUTLINE: This is a dose-escalation study of tagraxofusp in combination with azacitidine followed by a dose-expansion study.

Patients receive tagraxofusp intravenously (IV) over 15 minutes once daily (QD) on days 1-3 and azacitidine IV over 10-40 minutes QD on days 1-5 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and bone marrow aspiration and biopsy on study.

After completion of study treatment, patients are followed up at 30 days and then annually for up to 2 years after start of protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies.

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: 18-75 years old
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* First or second allogeneic HCT-eligible patients with AML or MDS with high-risk cytogenetics per European LeukemiaNet (ELN) (AML) or Revised International Prognostic Scoring System (R-IPSS) (MDS); or by having active (morphological) or minimal residual disease (MRD)+ status at the time of HCT (by multicolor flowcytometry, cytogenetics or molecular testing) OR patients who underwent HCT for AML or MDS with high-risk cytogenetics per ELN (AML) or R-IPSS (MDS)
* Positive for CD123 by flow cytometry of either peripheral blood or bone marrow aspirates at the time of diagnosis at any time-point prior to HCT. (Note: CD123 measurement will be conducted using the 10-color Beckman Coulter Navios XL flow cytometer. We will use CD123 PE [Beckman Coulter #A32535] to gate the abnormal population of interest. This population will be compared to the internal negative control population [e.g., T-cells]. If more than 20% of the abnormal population is positive relative to this control, it will be classified as positive.)
* Any conditioning regiment or GVHD prophylaxis is allowed
* Any donor (i.e., match related/unrelated, mismatched, haploidentical, etc.) or graft source (i.e., bone marrow, mobilized peripheral blood stem cells, etc.) is allowed
* Prior treatment with CD123-therapy is allowed if no progression is documented on therapy
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* STUDY MAINTENANCE TREATMENT: Complete response (CR) or MRD-positive on day 30 bone marrow biopsy (BMB) for disease assessment
* STUDY MAINTENANCE TREATMENT: Patients must be fully engrafted after HCT before starting the first cycle of maintenance. Full engraftment is defined as absolute neutrophil count (ANC) of 500 or above for 3 days and platelet count of more than 20,000 without transfusion for 7 consecutive days
* STUDY MAINTENANCE TREATMENT: ECOG ≤ 2
* STUDY MAINTENANCE TREATMENT: No treatment with anti-CD123 therapy after allogeneic HCT
* STUDY MAINTENANCE TREATMENT: No evidence of active or uncontrolled infection
* STUDY MAINTENANCE TREATMENT: No active GVHD; prednisone dose of ≤ 10 mg/daily is allowed
* STUDY MAINTENANCE TREATMENT: ANC ≥ 1.5 (within 7 days of day 1 of the cycle 1)

  * NOTE: Transfusion (red blood cells [RBC] or platelet) to achieve the above-mentioned counts is allowed
* STUDY MAINTENANCE TREATMENT: Hemoglobin (HbG) ≥ 7 (within 7 days of day 1 of the cycle 1)

  * NOTE: Transfusion (RBC or platelet) to achieve the above-mentioned counts is allowed
* STUDY MAINTENANCE TREATMENT: Platelet count ≥ 20K (within 7 days of day 1 of the cycle 1)

  * NOTE: Transfusion (RBC or platelet) to achieve the above-mentioned counts is allowed
* STUDY MAINTENANCE TREATMENT: Total bilirubin ≤ 2 x upper limit of normal (ULN) (unless has Gilbert's disease) (within 7 days of day 1 of the cycle 1)
* STUDY MAINTENANCE TREATMENT: Aspartate aminotransferase (AST) ≤ 2.5 x ULN (within 7 days of day 1 of the cycle 1)
* STUDY MAINTENANCE TREATMENT: Alanine aminotransferase (ALT) ≤ 2.5 x ULN (within 7 days of day 1 of the cycle 1)
* STUDY MAINTENANCE TREATMENT: Serum albumin > 3.2 (within 7 days of day 1 of the cycle 1) (note that albumin infusions are not permitted in order to enable eligibility but can be given after treatment starts)
* STUDY MAINTENANCE TREATMENT: Creatinine clearance of ≥ 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 7 days of day 1 of the cycle 1)
* STUDY MAINTENANCE TREATMENT: If not receiving anticoagulants: International normalized ratio (INR) or prothrombin (PT) ≤ 1.5 x ULN (within 7 days of day 1 of the cycle 1)

  * If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* STUDY MAINTENANCE TREATMENT: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 7 days of day 1 of the cycle 1)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* STUDY MAINTENANCE TREATMENT: The Patient should agree to use acceptable contraceptive methods for the duration of the time in the study, and to continue to use contraceptive methods for 6 months following the end of study therapy
* STUDY MAINTENANCE TREATMENT: The patient may not have persistent clinically significant toxicities grade ≥ 1 from previous therapies, including cytotoxic chemotherapy, targeted therapies, biological therapies, or immunotherapies, not readily controlled by supportive measures (excluding alopecia, nausea, and fatigue)
* STUDY MAINTENANCE TREATMENT: The patient has not received treatment with another investigational agent within 14 days of study entry
* STUDY MAINTENANCE TREATMENT: The patient does not have clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication)
* STUDY MAINTENANCE TREATMENT: The patient does not have uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study
* STUDY MAINTENANCE TREATMENT: The patient does not have known active or suspected central nervous system (CNS) disease. If suspected, CNS disease should be ruled out with relevant imaging and/or examination of cerebrospinal fluid
* STUDY MAINTENANCE TREATMENT: The patient does not have uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements
* STUDY MAINTENANCE TREATMENT: The patient does not have any condition which, in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents (tagraxofusp and azacitidine)
* Females only: Pregnant or breastfeeding
* Any other condition including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness, that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* The patient has an active malignancy and/or cancer history that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) with substantial potential for recurrence and/or ongoing active malignancy must be discussed with the sponsor before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ, cervical intraepithelial neoplasia, organ-confined prostate cancer with no evidence of progressive disease
* The patient has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication)
* The patient has uncontrolled, clinically significant pulmonary disease (e.g. chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study
* The patient has known active or suspected central nervous system (CNS) disease. If suspected, CNS disease should be ruled out with relevant imaging and/or examination of cerebrospinal fluid
* Active hepatitis B or C or HIV infection
* The patient has any condition which, in the opinion of the investigator, places the patient at an unacceptably high risk for toxicities
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. AEs will be recorded by type, severity, duration, and attribution or association with the study regimen and occurrence. Tables will be constructed to summarize the observed incidence, severity and type of toxicity. Point estimates and corresponding exact 95% confidence intervals (CIs) will be provided for each measure of toxicity/AEs.
Dose limiting toxicities (DLT) | Up to the end of cycle 1 on day 28
  DLTs will be graded according to the NCI CTCAE v5.0. AEs will be recorded by type, severity, duration, and attribution or association with the study regimen and occurrence. Tables will be constructed to summarize the observed incidence, severity and type of toxicity. Point estimates and corresponding exact 95% CIs will be provided for each measure of toxicity/AEs.
Percent of patients completing at least 3 cycles at assigned dose level | Up to 180 days
  Feasibility will be defined as 50% of patients completing at least 3 cycles of maintenance therapy at the assigned dose level. The point estimate and exact 95% CIs will be provided.

SECONDARY OUTCOMES:
Overall survival (OS) | From start of protocol therapy to death, assessed at 100 days and 1 year
  OS will be analyzed using the Kaplan-Meier curves.
Progression-free survival (PFS) | From start of protocol therapy to relapse or progression, or death, assessed at 100 days and 1 year
  PFS will be analyzed using the Kaplan-Meier curves.
Relapse/progression | From start of therapy to the first observation of relapse or progression, assessed at 100 days and 1 year
Non-relapse mortality | From start of therapy until non-disease related death, assessed at 100 days and 1 year
Incidence of grades 2-4 and 3-4 acute graft versus host disease (aGVHD) | From start of protocol therapy to aGVHD onset date, assessed up to 100 days
  AGVHD will be estimated using the cumulative incidence curve. AGVHD will be graded according to the Mount Sinai Acute Graft Versus Host Disease International Consortium Grading System.
Incidence of secondary graft failure | Up to 1 year post transplant
  Incidence of secondary graft failure will be defined as cytopenias after initial engraftment (absolute neutrophil count < 500/uL) with donor chimerism of less than 5% or falling donor chimerism with intervention such as second transplant or donor lymphocyte infusion or death due to cytopenias, and fall in donor chimerism, even if chimerism was > 5%.
Incidence of chronic graft versus host disease (cGVHD) | From start of protocol therapy to cGVHD onset date, assessed up to 1 year post transplant
  CGVHD will be scored according to National Institute of Health Consensus Staging. CGVHD will be estimated using the cumulative incidence curve.
Infection rate | In the first 100 days from the start of maintenance therapy
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Z Pourhassan, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States